CLINICAL TRIAL: NCT07202663
Title: A Single Center, Two-part, Double-blind, Randomized, Placebo-controlled, Dose-escalation, Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of BB-025 or Placebo, Alone and Following a Single Dose of BB-031, in Healthy Volunteers
Brief Title: Study of BB-025, Alone and After BB-031, in Healthy Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Basking Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BB-CLIN-102
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Pharmacodynamics; Pharmacokinetics; Healthy Volunteers
Keywords: Basking Biosciences; BB-025; BB-031; Reversal agent; Stroke; Acute Ischemic Stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: A randomized, placebo-controlled, double-blind, dose escalation to evaluate the safety, PK and PD of a single dose of investigational drug BB-025 or placebo, alone and following a single dose of BB-031, in healthy volunteers
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single Ascending Dose BB-025 (Experimental): Drug: BB-025, Investigational Drug
  Interventions: Drug: BB-025
- Single Dose Placebo (Placebo Comparator): Drug: Matched placebo to BB-025 cohorts
  Interventions: Drug: BB-025
- Single Dose BB-031 (Experimental): Drug: BB-031, Investigational Drug
  Interventions: Drug: BB-031

INTERVENTIONS:
Drug: BB-025 — Reversal agent for BB-031
  Arms: Single Ascending Dose BB-025; Single Dose Placebo
Drug: BB-031 — RNA aptamer
  Arms: Single Dose BB-031

SUMMARY:
The goal of this 2-part clinical trial is to learn about the safety and pharmacokinetics (PK) of a single dose of BB-025 when given on its own and after being given BB-031. Researchers will compare BB-025 to placebo (a look-alike substance that contains no drug) both on its own and after being given a single dose of BB-031 to assess the use of BB-025 as a reversal agent.

In the first part of the study, participants will receive a single dose of BB-025 or placebo. They will be followed for 28 days to check if they have any symptoms.

In the second part of the study, participants will receive a single dose of BB-031 and then be given either BB-025 or placebo. These participants will also be followed for 28 days to check if they have any symptoms.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years of age
* Ability to provide written consent
* Weight 50-100 kg with BMI 18-32 kg/m2
* Willingness to use contraceptives
* Negative results for alcohol and drugs of abuse

Exclusion Criteria:

* Pregnant or lactating females
* Familial bleeding disorder or individual or family history of bleeding diathesis or coagulopathy
* Females with active menstruation on day of dosing
* Use of prescription medications known to affect platelet function
* Use of NSAIDs, aspirin, anti-platelet or anti-coagulation therapy within 10 days of dosing
* Contraindication to anticoagulation or increased bleeding risks
* History of thrombocytosis, high platelet count, intracranial bleeding, aneurysm, stroke, vascular disease
* History of peptic ulcer disease, gastrointestinal or genitourinary bleed, severe trauma, fracture, major surgery of biopsy of parenchymal organ within past 3 months
* Planned surgery during the study
* Any clinically significant abnormality at screening
* Use of investigational drug in past 30 days or 5 half lives
* Concurrent enrollment in another clinical study or more than 4 clinical studies in past 12 months
* Any prior history of substance abuse or treatment or positive urine screen for drugs of abuse or positive breathalyzer test

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Safety as assessed by adverse events (AEs) | From dosing of study drug to final visit (Day 28)
  Incidence of treatment-emergent AEs

SECONDARY OUTCOMES:
Pharmacokinetics as measured by BB-025 plasma levels | From dosing to 24 hours after dosing
  Plasma concentrations of BB-025 (after single dose of drug)
Pharmacokinetics as measured by BB-031 plasma levels | From dosing to 24 hours after dosing
  Plasma concentrations of BB-031 (after single dose of drug)
Pharmacokinetics as measured by BB-025/BB-031 Complex plasma levels | From dosing of BB-031 through 24 hours after dosing of BB-025
  Plasma concentration of BB-025/BB-031 Complex after a single dose of each drug
Plasma von Willebrand Factor (vWF) Levels | From dosing of BB-031 or BB-025 to 24 hours after dosing of BB-025
  Level of vWF following administration of study drug
Platelet Function | From dosing of BB-031 or BB-025 to 24 hours after BB-025 dosing
  Whole blood platelet function closure times

CONTACTS AND LOCATIONS:
Overall Officials: Chris Argent, MD, Principal Investigator — Scientia Clinical Research Limited
Locations (1):
- Scintia Clinical Research Ltd, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No
Publication from this study not anticipated to need IPD data to be shared